CLINICAL TRIAL: NCT06639087
Title: Phase Ib Randomised, Placebo-controlled, Double-blind, Multicentre Study to Assess the Effects and Safety of AZD5462 on Top of Dapagliflozin in Participants With Heart Failure and Moderate Renal Impairment
Brief Title: A Phase Ib Study of AZD5462 on Top of Dapagliflozin in Participants With Heart Failure and Moderate Renal Impairment
Acronym: AURORA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D9090C00007; 2024-513142-11-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2024-09-13; First posted 2024-10-15 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Renal Impairment; Heart Failure
Keywords: Relaxin family peptide receptor 1 agonist; Estimated glomerular filtration rate; Heart failure; Renal impairment
MeSH Terms: conditions — Renal Insufficiency; Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD5462 + dapagliflozin (Active Comparator): Participants will receive AZD5462 on top of dapagliflozin once daily.
  Interventions: Drug: AZD5462; Drug: Dapagliflozin
- Placebo + dapagliflozin (Placebo Comparator): Participants will receive placebo on top of dapagliflozin once daily.
  Interventions: Drug: Dapagliflozin; Other: Placebo

INTERVENTIONS:
Drug: AZD5462 — Participants will receive AZD5462 on top of dapagliflozin once daily.
  Arms: AZD5462 + dapagliflozin
Drug: Dapagliflozin — Participants will receive dapagliflozin once daily with AZD5462 or placebo.
Other: Placebo — Participants will receive placebo on top of dapagliflozin once daily.
  Arms: Placebo + dapagliflozin

SUMMARY:
A study to investigate the effects and safety of AZD5462 on top of dapagliflozin in participants with heart failure and moderate renal impairment.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase 1b study to evaluate the safety, pharmacodynamics, and pharmacokinetics of AZD5462 on top of dapagliflozin in participants with heart failure and renal impairment.

The study will include 5 periods and approximately 9 study site visits:

* Screening Period of up to 4 weeks (at least one study visit)
* Run-in Period of up to 4 weeks (one study visit)
* Inpatient Treatment Period of 4 days (one study visit)
* Outpatient Treatment Period of up to 4 weeks (three study visits)
* Follow-up Period of up to 4 weeks (three study visits)

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a pre-existing diagnosis of heart failure (HF).
* Participants must have a left ventricular ejection fraction (LVEF) of ≤ 40% based on echocardiography taken within the last 9 months.
* Participants must have an estimated glomerular filtration rate (eGFR) of 30 to 60 milliliters per minute per 1.73 meters squared (mL/min/1.73 m2) (inclusive) at Screening as assessed by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) 2021 (creatinine) equation.
* Participants must be on stable HF standard of care (SoC) medication for at least 4 weeks prior to Screening. If the participant is currently taking diuretics, then diuretics must also be stable for at least one week prior to Screening.
* Participants must be on stable Sodium-glucose co-transporter-2 inhibitors (SGLT2) inhibitor treatment for at least 12 weeks prior to Screening.
* Minimum BMI of 18 kilograms per meter squared (kg/m2) at Screening.

Exclusion Criteria:

* Historical or current evidence of a clinically significant disease or disorder.
* Participants with a known hypersensitivity to AZD5462 or dapagliflozin, or to any of the excipients of these drug products.
* Congenital long QT syndrome or history of QT prolongation associated with other medications that required discontinuation of that medication.
* Cardiac ventricular arrhythmia that requires treatment. However, participants with atrial fibrillation or flutter and controlled ventricular rate (eg, resting heart rate < 110 beats per minute) are permitted. Participants with cardiac ventricular arrhythmia that are treated with antiarrhythmic agents (eg, amiodarone) and are stable are permitted.
* History of or anticipated heart transplant.
* Any planned highly invasive cardiovascular procedure (eg, coronary revascularisation, valve repair/replacement, aortic aneurysm surgery).
* Any evidence of clinically important disease or disorder which in the Investigator's opinion makes it undesirable for the participant to participate in the study.
* Positive hepatitis C antibody, hepatitis B virus surface antigen, or hepatitis B virus core antibody at Screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Change in sodium excretion | From Baseline to Day 1
  To evaluate the effect of AZD5462 on top of dapagliflozin in participants with heart failure (HF) and renal impairment.

SECONDARY OUTCOMES:
Change in urine albumin-creatinine ratio (uACR) | From Baseline to Day 1 and 29
  To evaluate the effect of AZD5462 on top of dapagliflozin in participants with HF and renal impairment.
Change in haematocrit | From Baseline to Day 29
  To evaluate the effect of AZD5462 on top of dapagliflozin in participants with HF and renal impairment.
Number of adverse events (AEs) and Serious Adverse Events (SAEs) | From Baseline to Day 57
  To evaluate the effect of AZD5462 on top of dapagliflozin in participants with HF and renal impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/